CLINICAL TRIAL: NCT04709133
Title: Clinical Outcomes Of Multi-ligament Knee Injuries In Assiut University Hospitals
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mohammed Abdelnasser Abdelfatah Farghay, Assistant lecturer at orthopedic and trauma department assiut university hospital, Assiut University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AssiutUMAAFMD
Record Dates: First submitted 2021-01-12; First posted 2021-01-14 (Actual); Last update posted 2021-01-14 (Actual); Status verified 2021-01

CONDITIONS: Knee Injuries
Keywords: Multi-ligament Knee Assiut Outcomes
MeSH Terms: conditions — Knee Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- multi-ligament knee injures (Experimental): A chart review will be performed to identify patients who underwent surgical treatment for multiligamentous knee injuries at Assiut University Hospital performed by one of sports medicine orthopaedic surgeons at Assiut arthroscopy and sport unit.
  Interventions: Procedure: multi-ligament knee surgery

INTERVENTIONS:
Procedure: multi-ligament knee surgery — a chart review will be performed to identify patients who underwent surgical treatment for multi-ligamentous knee injuries at Assiut University Hospital performed by one of sports medicine orthopaedic surgeons at Assiut arthroscopy and sport unit.

SUMMARY:
Multi-ligament knee injuries (MLKI) are devastating injuries. They are defined as injuries to at least two of the four major ligaments in the knee: anterior cruciate ligament, posterior cruciate ligament, lateral collateral ligament (and posterolateral corner) and medial collateral ligament (and posteromedial corner). These injuries are commonly classified using the Schenck classification system. The incidence of these injuries has been reported to be around 0.02-0.20% of all orthopaedic injuries. However, this is likely to be an underestimation due to spontaneous knee reduction and missed injuries. The immediate management of these injuries is crucial in identifying and treating any vascular and nerve injury. The literature has shown poor outcome and residual instability in those who were treated non-operatively. However, the optimal surgical treatment for these injuries is not known, with differences in opinion amongst treating clinicians. There are controversies in the timing of surgery (early versus delayed), single-staged or two-staged procedures and whether the damaged ligaments should be repaired or reconstructed

DETAILED DESCRIPTION:
Approximately 50% of all knee dislocations reduce spontaneously before the physician's arrival. Thus, high suspicion must be held, and literally every MLKI must be treated immediately as a true knee dislocation until proven otherwise. Failing to recognize the whole injury pattern around the knee can lead to disastrous consequences. Thus, an initial interdisciplinary systematic approach obtains top priority. Even though diagnostic image instruments become more and more reliable, physical examination still remains a fundamental element in any accurate assessment of knee dislocation. Several authors describe their own experiences and related treatment strategies of knee dislocation. But although a large number of studies about knee dislocation and MLKI do exist in medical databases, the complexity of this injury, the inhomogeneity of literature, and the persevering controversies in their treatment still make it difficult to draw reliable general conclusions.

Although important advances have been made in knee arthroscopy, ligament reconstruction and patient management, recommendations are not always applicable in settings with limited resources available. Challenges encountered in these situations include long delays to presentation, as well as the lack of sufficient access to operating room time, arthroscopic equipment, newer fixation devices, and allografts. Patients are often uninsured; work informally as manual laborers and their access to physiotherapy is very limited.

The purpose of this study is to analyse our institution's experience with multi-ligament knee injuries via the following items prevalence, detailed initial management at emergency department, types of these injuries, rationale of definitive treatment, rehabilitation protocol, postoperative complications and functional outcomes.

ELIGIBILITY:
Inclusion Criteria:

* • Patients presented to emergency department of Assiut University Hospital with knee dislocation.

  * Patients presented to outpatient sport clinics of Assiut University Hospital with two or more ligamentous knee injury.
  * Age from 18-55 years old.
  * Uninjured contralateral knee.
  * Informed consent obtained by the patient.

Exclusion Criteria:

* • Advanced knee osteoarthritis.

  * Current ipsilateral knee septic arthritis.
  * Patient with current psychological disease.
  * Patient with medically managed severe systemic disease.
  * Recent history of substance abuse (i.e. recreational drugs, alcohol) that would preclude reliable assessment.
  * Prisoner.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 4 (Estimated)
Dates: Start 2021-01 (Estimated); Primary Completion 2022-12 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
The arabic translated and validated Lysholm Knee Score | 6 months
  a chart review will be performed to identify patients who underwent surgical treatment for multiligamentous knee injuries at Assiut University Hospital performed by one of sports medicine orthopaedic surgeons at Assiut arthroscopy and sport unit.

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of medicine Assiut University, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Fanelli GC, Fanelli DG. Multiple Ligament Knee Injuries. J Knee Surg. 2018 May;31(5):399-409. doi: 10.1055/s-0038-1636910. Epub 2018 Mar 13. PMID 29534271